CLINICAL TRIAL: NCT00634049
Title: Open-label Study of Isavuconazole in the Treatment of Participants With Aspergillosis and Renal Impairment or of Participants With Invasive Fungal Disease Caused by Rare Moulds, Yeasts or Dimorphic Fungi
Brief Title: Isavuconazole in the Treatment of Renally Impaired Aspergillosis and Rare Fungi
Acronym: VITAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9766-CL-0103; WSA-CS-003 (Other: Basilea Protocol ID); 2006-005003-33 (EudraCT Number)
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Aspergillosis; Invasive Fungal Infections
Keywords: invasive fungal infections caused by rare molds, rare yeasts; BAL8557; Isavuconazole; Aspergillosis; or by dimorphic fungi; ASP9766
MeSH Terms: conditions — Aspergillosis; Invasive Fungal Infections | interventions — isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Isavuconazole (Experimental): Administration of isavuconazole 3 times a day in the vein (IV) or oral as a capsule for 2 days followed by daily administration of isavuconazole (IV) or oral
  Interventions: Drug: isavuconazole

INTERVENTIONS:
Drug: isavuconazole — Administration of 200 mg isavuconazole 3 times a day in the vein (IV) or oral as a capsule for 2 days, followed by daily administration of 200 mg isavuconazole (IV) or oral
  Other Names: BAL8557; ASP9766

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of isavuconazole in the treatment of renally impaired participants with invasive fungal infections caused by Aspergillus and participants with invasive fungal disease caused by rare fungi.

DETAILED DESCRIPTION:
Acute invasive fungal infections caused by aspergillus, rare moulds, yeasts or dimorphic fungi are life threatening diseases. Early treatment with highly effective anti-fungals reduces mortality. This study investigates the safety and efficacy of isavuconazole in participants with aspergillosis and renal impairment, and in participants suffering from invasive infections from rare fungi.

ELIGIBILITY:
Inclusion Criteria:

•Participants meeting EORTC/MSG (European Organization for the Research and Treatment of Cancer/Mycoses Study Group) definition of proven or culture positive probable IFD (invasive fungal disease) caused by rare moulds, yeasts, or dimorphic fungi (i.e. fungal pathogens other than Aspergillus fumigatus or Candida species) whether renally impaired or not (including dialysis) who require primary therapy for their IFD at the time of enrollment.

OR

•Participants who had proven or probable zygomycosis, whether renally impaired or not (including dialysis), who require primary therapy. Zygomycosis must be documented by culture or histology / cytology.

OR

•Participants meeting EORTC/MSG definition of proven or culture positive probable IFD caused by rare moulds, yeasts, or dimorphic fungi (i.e., fungal pathogens other than Aspergillus fumigatus or Candida species), whether RI or not (including dialysis), who were refractory to current treatment defined as,

* Clear documentation of progression of disease. Note: radiological progression only in association with white blood cell (WBC) count recovery was not acceptable.
* Failure to improve clinically despite receiving at least 7 days of standard antifungal regimen. Prior to enrolling patients who fell into this category, the Medical Monitor was contacted for approval.

OR

• Participants meeting EORTC/MSG definition of proven or culture positive probable IFD caused by rare moulds, yeasts, or dimorphic fungi (i.e., fungal pathogens other than Aspergillus fumigatus or Candida species), whether RI or not (including dialysis), who were intolerant to current treatment for example:

* Doubling of serum creatinine value to higher than the upper limit of normal (ULN) within 48 hours.
* Serum creatinine > 2.0 mg/mL and current treatment with polyene or IV voriconazole.
* Other significant drug-related adverse reaction(s) to the current antifungal agent, resulting in discontinuation of the treatment, e.g., persistence of visual disturbance, allergic reaction, phototoxicity or severe infusion reaction (hypertensive crisis, severe chills or shock).
* Documented inability to achieve adequate blood levels of posaconazole, voriconazole or itraconazole.

Exclusion Criteria:

* A known condition of the participants that may jeopardize adherence to the protocol requirements
* Participants who are unlikely to survive 30 days
* Participants with a body weight < 40 kg
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2008-04-22 (Actual); Primary Completion 2014-01-03 (Actual); Study Completion 2016-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (96):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City Of Hope National Medical Center, Duarte, California
  - University of California Davis Health System, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - University of California at San Francisco, San Francisco, California
  - Stanford University Hospital, Stanford, California
  - University Of Colorado Health Sciences Center, Aurora, Colorado
  - Emory Hospital, Atlanta, Georgia
  - University of Chicago, Division of Infectious Diseases, Chicago, Illinois
  - Indiana BMT, Beech Grove, Indiana
  - Infectious Disease of Indiana, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Brigham & Womens Hospital, Boston, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Wayne State University School of Medicine, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Upstate Infectious Diseases Association LLP, Albany, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Regional Infection Diseases Infusion Center Inc., Lima, Ohio
  - Temple University Health Sciences, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Clinical Research, Seattle, Washington
- Argentina (5):
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma
  - Hospital Nuestra Senora de la Misericordia, Córdoba
  - Hospital San Roque, Córdoba
  - Centro Polivalente de Asistencia e Investigación Clínica - CER San Juan, San Juan
- Australia (2):
  - Mater Medical Centre, South Brisbane
  - Princess Alexandria Hospital, Woolloongabba
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Erasme Hospital, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
- Brazil (7):
  - Hospital Felicio Rocho, Belo Horizonte
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Hospital das Clinicas da UFPR, Curitiba
  - Hospital de Clinicas da FMUSP - Ribeirao Preto, Ribeirão Preto
  - Hospital Universitario Clementino Fraga Filho, Rio de Janeiro
  - Hospital Universitario de Santa Maria, Santa Maria
  - Hospital Professor Edmundo Vasconcelos, São Paulo
- Canada (3):
  - Hamilton Health Sciences - Henderson Site, Hamilton, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Hôpital Maisonneuve - Rosemont, Montreal, Quebec
- Hospital Clinico San Borja Arriaran, Santiago, Chile
- Egypt (3):
  - Alexandria University Hospital, Alexandria
  - National Cancer Institute, Cairo
  - Nasser Institute, Cairo
- France (6):
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli Calmette - Marseille, Marseille
  - Hotel Dieu, Nantes
  - Hôpital Saint-Louis, Paris
  - Hopital Hautepierre, Strasbourg
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (5):
  - Universitaetsklinikum Aachen, Aachen
  - Charite-Campus Benjamin Franklin, Berlin
  - Universitaet Koeln, Cologne
  - Klinikum Neuperlach, München
  - Medizinische Klinik und Polyklinik II, Würzburg
- India (8):
  - Medanta Medicity Hospital, Gūrgaon, Haryan
  - Shirdi Sai Baba Cancer Hospital K. M. C. Hospital, Manipal, Kama
  - Tata Memorial Hopital, Department of Anesthesia, Mumbai, Mahara
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Mahara
  - Global Hospitals & Health City, Chennai, Tamilna
  - Sterling Hospital, Ahmedabad
  - Apollo Hospitals, Hyderabad
  - Sahyadri Specialty Hospital, Pune
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah Universtiy Hospital - Ein Kerem, Jerusalem
  - Rabin MC, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky MC Ichilov Hospital Tel Aviv, Tel Aviv
- Lebanon (3):
  - American University of Beirut Medical Center, Beirut
  - Clinique Dr. Rizk, Beirut
  - Rafik Hariri University Hospital, Beirut
- Mexico (4):
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador, Mexico City
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Hospital Central Dr Ignacio Morones Prieto, San Luis Potosí City
- Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw, Poland
- Russia (4):
  - S.I. Russian Oncological Research Center n.a. N.N. Blokhin, Moscow
  - State Institution "Hematology Research Center" RAMS, Moscow
  - Republican Hospital named after V.A. Baranov, Petrozavodsk
  - St-Petersburg MA Postgraduate Education, Saint Petersburg
- Private Practice, Lyttleton, Gauteng, South Africa
- South Korea (5):
  - Soonchunhyang University Bucheon Hospital, Buchon-si
  - Gachon University Gil Hospital, Incheon
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul
  - Asan Medical Center, Seoul
- Thailand (5):
  - Songklanagarind Hospital, Hat Yai
  - Maharat Nakhon Ratchasima Hospital, Muang
  - Srinagarind Hospital, Muang
  - Maharaj Nakorn Chiang Mai Hospital, Muang
  - Ramathibodi Hospital, Ratchathewi

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Hamed K, Engelhardt M, Kovanda LL, Huang JJ, Yan J, Aram JA. Post-hoc analysis of the safety and efficacy of isavuconazole in older patients with invasive fungal disease from the VITAL and SECURE studies. Sci Rep. 2023 Apr 25;13(1):6730. doi: 10.1038/s41598-023-31788-1. PMID 37185921
- [Derived] Kovanda LL, Desai AV, Lu Q, Townsend RW, Akhtar S, Bonate P, Hope WW. Isavuconazole Population Pharmacokinetic Analysis Using Nonparametric Estimation in Patients with Invasive Fungal Disease (Results from the VITAL Study). Antimicrob Agents Chemother. 2016 Jul 22;60(8):4568-76. doi: 10.1128/AAC.00514-16. Print 2016 Aug. PMID 27185799
- [Derived] Thompson GR 3rd, Rendon A, Ribeiro Dos Santos R, Queiroz-Telles F, Ostrosky-Zeichner L, Azie N, Maher R, Lee M, Kovanda L, Engelhardt M, Vazquez JA, Cornely OA, Perfect JR. Isavuconazole Treatment of Cryptococcosis and Dimorphic Mycoses. Clin Infect Dis. 2016 Aug 1;63(3):356-62. doi: 10.1093/cid/ciw305. Epub 2016 May 11. PMID 27169478
- [Derived] Marty FM, Ostrosky-Zeichner L, Cornely OA, Mullane KM, Perfect JR, Thompson GR 3rd, Alangaden GJ, Brown JM, Fredricks DN, Heinz WJ, Herbrecht R, Klimko N, Klyasova G, Maertens JA, Melinkeri SR, Oren I, Pappas PG, Racil Z, Rahav G, Santos R, Schwartz S, Vehreschild JJ, Young JH, Chetchotisakd P, Jaruratanasirikul S, Kanj SS, Engelhardt M, Kaufhold A, Ito M, Lee M, Sasse C, Maher RM, Zeiher B, Vehreschild MJGT; VITAL and FungiScope Mucormycosis Investigators. Isavuconazole treatment for mucormycosis: a single-arm open-label trial and case-control analysis. Lancet Infect Dis. 2016 Jul;16(7):828-837. doi: 10.1016/S1473-3099(16)00071-2. Epub 2016 Mar 9. PMID 26969258
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=51

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consenting adult participants with proven, probable or possible invasive aspergillosis and renally impaired (RI) or of participants with invasive fungal disease (IFD) caused by rare moulds, yeasts or dimorphic fungi meeting the inclusion and none of the exclusion criteria were considered for entry into the study.
Pre-assignment Details: Analysis and interpretation of the results was pathogen dependent and each pathogen was quite rare, therefore it was not feasible to enroll a sufficient number of participants in a randomized controlled trial to power the study adequately to allow statistical comparisons.
Groups:
- Isavuconazole: Participants received a loading dose of isavuconazole, 200 mg three times a day administered intravenously (IV) or orally (PO) [or per os (PO)] for the first 2 days followed by a maintenance dose from Day 3 of 200 mg once daily either IV or orally until they reached a treatment endpoint or for a maximum of 180 days; with an option for extended treatment under specified criteria.
Period: Overall Study
Arm/Group | Isavuconazole
Started | 149
Completed | 146
Not Completed | 3
Not completed — Never received study drug | 1
Not completed — Died prior to receiving study drug | 1
Not completed — Screening failure | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population (ITT)
Arm/Group | Isavuconazole
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (16.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 108
  More than one race | 0
  Unknown or Not Reported | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 124
Region of Enrollment [Number; unit: participants]
  Brazil | 20
  India | 5
  Israel | 21
  Lebanon | 1
  Mexico | 8
  Russian Federation | 2
  Korea, Republic of | 2
  Thailand | 14
  Belgium | 13
  Germany | 4
  United States | 56
Therapy status [Number; unit: participants]
  Primary Therapy | 93
  Refractory | 38
  Intolerant | 12
  Missing | 3
Hematologic malignancy [Number; unit: participants]
  Yes | 63
  No | 83
Allogeneic Bone Marrow Transplant (BMT)/Hematopoietic Stem Cell Transplant (HSCT) [Number; unit: participants] — Allogeneic BMT/HSCT status was defined as yes for participants who noted allogeneic for type of transplant and bone marrow cells for type of cells on the primary underlying disease or condition electronic case report form (eCRF). Otherwise, allogeneic BMT/HSCT status equaled no.
  participants
    Yes | 26
    No | 120
Uncontrolled malignancy [Number; unit: participants] — Uncontrolled malignancy status was defined as yes for participants who noted a malignancy for diagnosis and new diagnosis/active disease or relapse for present status on the primary underlying disease or condition eCRF. Otherwise, uncontrolled malignancy status equaled no.
  participants
    Yes | 46
    No | 100
Neutropenic [Number; unit: participants] — Baseline neutropenic status was defined as yes for patients who noted recently resolved or ongoing neutropenia among the list of host factors on the categorization of IFD eCRF. Baseline neutropenic status was defined as no for patients who completed the categorization of IFD eCRF and did not meet the criterion in the previous sentence. Otherwise, baseline neutropenic status was missing.
  participants
    Yes | 38
    No | 66
    Missing | 42
Corticosteroid use [Number; unit: participants] — Corticosteroid use was defined as yes for participants who were administered corticosteroids for 21 days out of 28 days leading up to first administration of study drug. Otherwise, corticosteroid use equaled no.
  participants
    Yes | 35
    No | 111
T-cell immunosuppressant use [Number; unit: participants] — T-cell immunosuppressant use was defined as yes for patients who noted treatment with other recognized T-cell immunosuppressants among the list of host factors on the categorization of IFD eCRF. Along with the investigators' assessment, participants who took certain prior medications could have been considered based on the medical evaluation. T-cell immunosuppressant use was defined as no for participants who completed the categorization of IFD eCRF and did not meet the criterion in the previous sentences. Otherwise, T-cell immunosuppressant use was missing.
  participants
    Yes | 61
    No | 48
    Missing | 37

OUTCOME MEASURES:

1. Primary Outcome: Crude Success Rate of Overall Outcome of Treatment Evaluated by the Data Review Committee (DRC) at Day 42, 84 and End of Treatment (EOT).
Description: The DRC assessed overall response based on individual clinical, mycological and radiological response assessments. Overall response outcomes were described as Success (complete or partial). Complete success was defined as a resolution of all clinical symptoms and physical findings associated with IFD. Partial success was defined as a resolution of at least some clinical symptoms and physical findings associated with IFD End of treatment (EOT) is the last day of study drug administration, with an estimated duration up to 180 days.
Time Frame: Day 42, 84 and End of Treatment (EOT [Day 180])
Population: Modified Intent-To-Treat population (mITT)
Measure: Number; unit: percentage of participants
Groups:
- mITT - Aspergillus [Renally Impaired]: Aspergillus - Renally Impaired (RI) mITT population consisted of participants who have had proven or probable IFD as determined by the DRC. Classification by the DRC was based on the type of pathogen which was found to be the cause of participant's IFD. The Aspergillus-mITT population was presented by renal status, and whether they are renally impaired and not renally impaired. Renal impairment was defined as yes for participants who had a baseline estimated glomerular filtration rate (eGFR-MDRD) < 60 mL/min/1.73 m^2, no for patients who had a baseline eGFR-MDRD ≥ 60 mL/min/1.73 m^2. Overall there were 24 participants in the mITT-Aspergillus population out of which 20 participants were classified as Renally Impaired (RI).
- mITT - Aspergillus [Not Renally Impaired]: Aspergillus - Not Renally Impaired (NRI) mITT population consisted of participants who had proven or probable IFD as determined by the DRC. Classification by the DRC was based on the type of pathogen which was found to be the cause of participant's IFD. The Aspergillus-mITT population was presented by renal status (Renally Impaired and Not Renally Impaired). Overall there were 24 participants in the mITT- Aspergillus population out of which 4 participants were classified as Not Renally Impaired (NRI).
- mITT - Mucorales (Primary Therapy): Mucorales - Primary Therapy mITT population consisted of participants who had proven or probable IFD as determined by the DRC. Based on the DRC assessment 37 participants were assessed proven or probable Mucorales infection (32 participants had proven and 5 participants had probable invasive mucormycosis). The DRC also categorized each patient by therapy status; these groups were primary therapy, refractory and intolerant. There were 21 participants receiving isavuconazole as a primary therapy.
- mITT - Mucorales (Refractory): Mucorales - Refractory Therapy mITT population consisted of participants who had proven or probable IFD as determined by the DRC. Based on the DRC assessment 37 participants were assessed to have proven or probable Mucorales infection (32 participants had proven and 5 participants had probable invasive mucormycosis).The DRC also categorized each participant by therapy status; these groups were primary therapy, refractory and intolerant. There were 11 participants whose IFD was refractory to prior antifungal therapy (AFT)
- mITT - Mucorales (Intolerant): Mucorales - Intolerant mITT population consisted of participants who had proven or probable IFD as determined by the DRC. Based on the DRC assessment 37 participants were assessed to have proven or probable Mucorales infection (32 participant had proven and 5 participants had probable invasive mucormycosis). The DRC also categorized each participant by therapy status; these groups were primary therapy, refractory and intolerant. There were 5 participants who were intolerant to prior antifungal therapy (AFT).
- mITT- Other Filamentous Fungi: Other Filamentous Fungi mITT population consisted of 17 participants who had proven or probable IFD as determined by the DRC caused by other filamentous fungi (4 Fusarium, 2 Exophiala, 2 Cladosporium, 2 Scopulariopsis and 1 each of Acremonium, Alternaria, Curvularia, Exserohilum, Paecilomyces, Pseudallescheria and Scedosporium).
- mITT- Other Mould Species Only: Other Mould Species mITT population consisted of 7 participants who had proven or probable IFD as determined by the DRC caused by mould species.
- mITT- Other Dimorphic Fungi: Other Dimorphic Fungi mITT population consisted of 29 participants who had proven or probable IFD as determined by the DRC caused by dimorphic fungi (10 Paracoccidiodes, 9 Coccidiodides, 7 Histoplasma, 3 Blastomyces).
- mITT- Other Non-Candida Yeast: Other non-Candida Yeast mITT population consisted of 11 participants who had proven or probable IFD as determined by the DRC caused by non-Candida yeast (4 Cryptococcus neoformans, 3 Cryptococcus gatii, 2 Cryptococcus not otherwise specified (NOS) and 2 Trichosporon).
- mITT-Other Mixed Infection: Other Mixed Infections mITT group consisted of 15 participants who had proven or probable IFD as determined by the DRC caused by mixed infections aspergillosis/mucormycosis.
Arm/Group | mITT - Aspergillus [Renally Impaired] | mITT - Aspergillus [Not Renally Impaired] | mITT - Mucorales (Primary Therapy) | mITT - Mucorales (Refractory) | mITT - Mucorales (Intolerant) | mITT- Other Filamentous Fungi | mITT- Other Mould Species Only | mITT- Other Dimorphic Fungi | mITT- Other Non-Candida Yeast | mITT-Other Mixed Infection
Number analyzed (Participants) | 20 | 4 | 21 | 11 | 5 | 17 | 7 | 29 | 11 | 15
percentage of participants
  Day 42- Success Rate | 25.0 | 50.0 | 14.3 | 9.1 | 0 | 47.1 | 28.6 | 41.4 | 36.4 | 13.3
  Day 84 - Success Rate | 30.0 | 25.0 | 9.5 | 36.4 | 20.0 | 41.2 | 28.6 | 44.8 | 36.4 | 13.3
  End of Treatment (EOT) - Success Rate | 30.0 | 66.7 | 31.6 | 36.4 | 20.0 | 64.7 | 28.6 | 64.3 | 72.7 | 14.3

2. Secondary Outcome: Crude Success Rate of Clinical Response to Treatment Evaluated by the Data Review Committee (DRC) at Day 42, 84 and EOT
Description: The DRC evaluated clinical response to treatment at day 42, day 84 and EOT. Clinical response outcomes were described as Success [Resolution of all attributable clinical symptoms and physical findings and Partial resolution of attributable clinical symptoms and physical findings]. End of treatment (EOT) is the last day of study drug administration, with an estimated duration up to 180 days.
Time Frame: Day 42, 84 and End of Treatment (EOT [Day 180])
Population: Modified Intent-To-Treat population (mITT)
Measure: Number; unit: percentage of participants
Groups:
- mITT - Aspergillus [Renally Impaired]: Aspergillus - Renally Impaired (RI) mITT population consisted of participants who have had proven or probable IFD as determined by the DRC. Classification by the DRC was based on the type of pathogen which was found to be the cause of participant's IFD. The Aspergillus-mITT population was presented by renal status, and whether they are renally impaired or not renally impaired. Renal impairment was defined as yes for participants who had a baseline estimated glomerular filtration rate (eGFR-MDRD) < 60 mL/min/1.73 m^2, no for patients who had a baseline eGFR-MDRD ≥ 60 mL/min/1.73 m^2. Overall there were 24 participants in the mITT-Aspergillus population out of which 20 participants were classified as Renally Impaired (RI).
- mITT - Mucorales (Refractory): Mucorales - Refractory Therapy mITT population consisted of participants who had proven or probable IFD as determined by the DRC. Based on the DRC assessment 37 participants were assessed to have proven or probable Mucorales infection (32 participants had proven and 5 participants had probable invasive mucormycosis).The DRC also categorized each patient by therapy status; these groups were primary therapy, refractory and intolerant. There were 11 participants whose IFD was refractory to prior AFT.
- mITT - Mucorales (Intolerant): Mucorales - Intolerant mITT population consisted of participants who had proven or probable IFD as determined by the DRC. Based on the DRC assessment 37 participants were assessed to have proven or probable Mucorales infection (32 participant had proven and 5 participants had probable invasive mucormycosis). The DRC also categorized each participant by therapy status; these groups were primary therapy, refractory and intolerant. There were 5 participants who were intolerant to prior AFT.
- mITT-Other Filamentous Fungi: Other Filamentous Fungi mITT population consisted of 17 participants who had proven or probable IFD as determined by the DRC caused by other filamentous fungi (4 Fusarium, 2 Exophiala, 2 Cladosporium, 2 Scopulariopsis and 1 each of Acremonium, Alternaria, Curvularia, Exserohilum, Paecilomyces, Pseudallescheria and Scedosporium).
- mITT- Other Mould Species Only: Other Mould Species mITT population consisted of 7 participants who have had proven or probable IFD as determined by the DRC caused by mould species.
Arm/Group | mITT - Aspergillus [Renally Impaired] | mITT - Aspergillus [Not Renally Impaired] | mITT - Mucorales (Primary Therapy) | mITT - Mucorales (Refractory) | mITT - Mucorales (Intolerant) | mITT-Other Filamentous Fungi | mITT- Other Mould Species Only | mITT- Other Dimorphic Fungi | mITT- Other Non-Candida Yeast | mITT-Other Mixed Infection
Number analyzed (Participants) | 20 | 4 | 21 | 11 | 5 | 17 | 7 | 29 | 11 | 15
percentage of participants
  Day 42- Success Rate | 55.0 | 75.0 | 50.0 | 33.3 | 50.0 | 68.8 | 71.4 | 79.3 | 70.0 | 42.9
  Day 84 - Success Rate | 45.0 | 25.0 | 40.0 | 22.2 | 50.0 | 62.5 | 42.9 | 82.8 | 70.0 | 35.7
  End of Treatment (EOT) - Success Rate | 55.0 | 66.7 | 55.6 | 22.2 | 50.0 | 81.3 | 85.7 | 82.1 | 70.0 | 38.5

3. Secondary Outcome: Crude Success Rate of Mycological Response to Treatment Evaluated by the Data Review Committee (DRC) at Day 42, 84 and EOT
Description: The DRC evaluated mycological response to treatment at day 42, day 84 and EOT. Mycological response outcomes were described as Success [Eradication and Presumed eradication]. End of treatment (EOT) is the last day of study drug administration, with an estimated duration up to 180 days.
Time Frame: Day 42, 84 and End of Treatment (EOT [Day 180])
Population: Modified Intent-To-Treat population (mITT)
Measure: Number; unit: percentage of participants
Groups:
- mITT - Aspergillus [Renally Impaired]: Aspergillus - Renally Impaired mITT population consisted of participants who have had proven or probable IFD as determined by the DRC. Classification by the DRC was based on the type of pathogen which was found to be the cause of participants IFD. The Aspergillus-mITT population was presented by renal status, renally impaired and not renally impaired. Renal impairment was defined as yes for participants who have a baseline estimated glomerular filtration rate (eGFR-MDRD) < 60 mL/min/1.73 m^2, no for participants who have a baseline eGFR-MDRD ≥ 60 mL/min/1.73 m^2. Overall there were 24 participants in the mITT-Aspergillus population out of which 20 participants were classified as Renally Impaired (RI).
- mITT-Other Mixed Infection: Other Mixed Infections mITT population consisted of 15 participants who have had proven or probable IFD as determined by the DRC caused by mixed infections aspergillosis/mucormycosis.
Arm/Group | mITT - Aspergillus [Renally Impaired] | mITT - Aspergillus [Not Renally Impaired] | mITT - Mucorales (Primary Therapy) | mITT - Mucorales (Refractory) | mITT - Mucorales (Intolerant) | mITT-Other Filamentous Fungi | mITT- Other Mould Species Only | mITT- Other Dimorphic Fungi | mITT- Other Non-Candida Yeast | mITT-Other Mixed Infection
Number analyzed (Participants) | 20 | 4 | 21 | 11 | 5 | 17 | 7 | 29 | 11 | 15
percentage of participants
  Day 42- Success Rate | 30.0 | 50.0 | 4.8 | 0 | 0 | 29.4 | 28.6 | 27.6 | 45.5 | 13.3
  Day 84 - Success Rate | 35.0 | 25.0 | 9.5 | 27.3 | 40.0 | 35.3 | 28.6 | 27.6 | 45.5 | 13.3
  End of Treatment (EOT) - Success Rate | 35.0 | 66.7 | 31.6 | 36.4 | 40.0 | 70.6 | 28.6 | 53.6 | 81.8 | 14.3

4. Secondary Outcome: Crude Success Rate of Radiological Response to Treatment Evaluated by the Data Review Committee (DRC) at Day 42, 84 and EOT
Description: The DRC evaluated radiological response to treatment at at day 42, day 84 and EOT. Radiological response outcomes were described as Success [Improvement of at least 25% from baseline for invasive aspergillosis and other filamentous mold infections], [Improvement of at least 50% from baseline for invasive aspergillosis and other filamentous mold infections]; and [Improvement of at least 25% from baseline if EOT occurs prior to day 42 and at least 50% improvement from baseline if EOT occurs after day 42 for invasive aspergillosis and other filamentous mold infections]. End of treatment (EOT) is the last day of study drug administration, with an estimated duration up to 180 days.
Time Frame: Day 42, 84 and End of Treatment (EOT [Day 180])
Population: Modified Intent-To-Treat population (mITT)
Measure: Number; unit: percentage of participants
Groups:
- mITT - Aspergillus [Not Renally Impaired]: Aspergillus - Renally Impaired mITT population consisted of participants who have had proven or probable IFD as determined by the DRC. Classification by the DRC was based on the type of pathogen which was found to be the cause of participants IFD. The Aspergillus-mITT population was presented by renal status, renally impaired and not renally impaired. Overall there were 24 participants in the mITTAspergillus population out of which 4 participants were classified as Not Renally Impaired (NRI).
- mITT - Mucorales (Primary Therapy): Mucorales - Primary Therapy mITT population consisted of participants who have had proven or probable IFD as determined by the DRC. Based on the DRC assessment 37 participants were assessed to have proven or probable Mucorales infection (32 participants had proven and 5 participants had probable invasive mucormycosis). The DRC also categorized each patient by therapy status; these groups were primary therapy, refractory and intolerant. There were 21 participants receiving isavuconazole as a primary therapy.
- mITT - Mucorales (Refractory): Mucorales - Refractory Therapy mITT population consisted of participants who have had proven or probable IFD as determined by the DRC. Based on the DRC assessment 37 participants were assessed to have proven or probable Mucorales infection (32 participants had proven and 5 participants had probable invasive mucormycosis).The DRC also categorized each patient by therapy status; these groups were primary therapy, refractory and intolerant. There were 11 participants whose IFD was refractory to prior AFT.
- mITT - Mucorales (Intolerant): Mucorales - Intolerant mITT population consisted of participants who have had proven or probable IFD as determined by the DRC. Based on the DRC assessment 37 participants were assessed to have proven or probable Mucorales infection (32 participant had proven and 5 participants had probable invasive mucormycosis). The DRC also categorized each participant by therapy status; these groups were primary therapy, refractory and intolerant. There were 5 participants who were intolerant to prior AFT.
- mITT-Other Filamentous Fungi: Other Filamentous Fungi mITT population consisted of 17 participants who have had proven or probable IFD as determined by the DRC caused by other filamentous fungi (4 Fusarium,2 Exophiala,2 Cladosporium,2 Scopulariopsis and 1 each of Acremonium, Alternaria, Curvularia,Exserohilum, Paecilomyces,Pseudallescheria and Scedosporium).
- mITT- Other Dimorphic Fungi: Other Dimorphic Fungi mITT population consisted of 29 participants who have had proven or probable IFD as determined by the DRC caused by dimorphic fungi (10 Paracoccidiodes,9 Coccidiodides, 7 Histoplasma, 3 Blastomyces).
- mITT- Other Non-Candida Yeast: Other Non Candida Yeast mITT population consisted of 11 participants who have had proven or probable IFD as determined by the DRC caused by non-Candida yeast (4 Cryptococcus neoformans, 3 Cryptococcus gatii, 2 Cryptococcus NOS and 2 Trichosporon).
Arm/Group | mITT - Aspergillus [Renally Impaired] | mITT - Aspergillus [Not Renally Impaired] | mITT - Mucorales (Primary Therapy) | mITT - Mucorales (Refractory) | mITT - Mucorales (Intolerant) | mITT-Other Filamentous Fungi | mITT- Other Mould Species Only | mITT- Other Dimorphic Fungi | mITT- Other Non-Candida Yeast | mITT-Other Mixed Infection
Number analyzed (Participants) | 20 | 4 | 21 | 11 | 5 | 17 | 7 | 29 | 11 | 15
percentage of participants
  Day 42- Success Rate | 30.0 | 25.0 | 0 | 10.0 | 0 | 25.0 | 16.7 | 21.4 | 0 | 7.1
  Day 84 - Success Rate | 20.0 | 25.0 | 4.8 | 20.0 | 20.0 | 6.3 | 0 | 28.6 | 10.0 | 14.3
  End of Treatment (EOT) - Success Rate | 15.0 | 66.7 | 16.7 | 20.0 | 20.0 | 50.0 | 0 | 33.3 | 10.0 | 7.7

5. Secondary Outcome: Crude Success Rate of Clinical Response to Treatment Evaluated by the Investigator at Day 42, Day 84 and EOT
Description: The Investigator evaluated clinical response to treatment at day 42, day 84 and EOT. Clinical response outcomes were described as Success [Resolution of all attributable clinical symptoms and physical findings] and [Resolution of some attributable clinical symptoms and physical findings]. End of treatment (EOT) is the last day of study drug administration, with an estimated duration up to 180 days.
Time Frame: Day 42, Day 84 and End of Treatment (EOT [Day 180])
Population: Modified Intent-To-Treat population (mITT)
Measure: Number; unit: percentage of participants
Groups:
- mITT - Aspergillus [Renally Impaired]: Aspergillus - Renally Impaired (RI) mITT population consisted of participants who have had proven or probable IFD as determined by the DRC. Classification by the DRC was based on the type of pathogen which was found to be the cause of participant's IFD. The Aspergillus-mITT population was presented by renal status, and whether they are renally impaired and not renally impaired. Renal impairment was defined as yes for participants who had a baseline estimated glomerular filtration rate (eGFR-MDRD) < 60 mL/min/1.73 m^2, no for participants who had a baseline eGFR-MDRD ≥ 60 mL/min/1.73 m^2. Overall there were 24 participants in the mITT-Aspergillus population out of which 20 participants were classified as Renally Impaired (RI).
Arm/Group | mITT - Aspergillus [Renally Impaired] | mITT - Aspergillus [Not Renally Impaired] | mITT - Mucorales (Primary Therapy) | mITT - Mucorales (Refractory) | mITT - Mucorales (Intolerant) | mITT- Other Filamentous Fungi | mITT- Other Mould Species Only | mITT- Other Dimorphic Fungi | mITT- Other Non-Candida Yeast | mITT-Other Mixed Infection
Number analyzed (Participants) | 20 | 4 | 21 | 11 | 5 | 17 | 7 | 29 | 11 | 15
percentage of participants
  Day 42 | 60.0 | 75.0 | 50.0 | 28.6 | 25.0 | 81.3 | 85.7 | 75.9 | 70.0 | 50.0
  Day 84 | 55.0 | 55.0 | 21.4 | 25.0 | 20.0 | 62.5 | 42.9 | 82.2 | 70.0 | 35.7
  End of Treatment (EOT) | 60.0 | 75.0 | 42.9 | 28.6 | 66.7 | 81.3 | 71.4 | 79.3 | 70.0 | 42.9

6. Secondary Outcome: Crude Success Rate of Mycological Response to Treatment Evaluated by the Investigator at Day 42, Day 84 and EOT
Description: The Investigator evaluated mycological response to treatment at day 42, day 84 and EOT. Mycological response outcomes were described as Success [Eradication,Presumed eradication]. End of treatment (EOT) is the last day of study drug administration, with an estimated duration up to 180 days.
Time Frame: Day 42, Day 84 and End of Treatment (EOT [Day 180])
Population: Modified Intent-To-Treat population (mITT)
Measure: Number; unit: percentage of participants
Arm/Group | mITT - Aspergillus [Renally Impaired] | mITT - Aspergillus [Not Renally Impaired] | mITT - Mucorales (Primary Therapy) | mITT - Mucorales (Refractory) | mITT - Mucorales (Intolerant) | mITT- Other Filamentous Fungi | mITT- Other Mould Species Only | mITT- Other Dimorphic Fungi | mITT- Other Non-Candida Yeast | mITT-Other Mixed Infection
Number analyzed (Participants) | 20 | 4 | 21 | 11 | 2 | 17 | 7 | 29 | 11 | 15
percentage of participants
  Day 42 | 46.7 | 66.7 | 50.0 | 28.6 | 25.0 | 69.2 | 83.3 | 70.6 | 50.0 | 18.2
  Day 84 | 44.4 | 50.0 | 21.4 | 25.0 | 20.0 | 64.3 | 42.9 | 80.0 | 25.0 | 33.3
  End of Treatment (EOT) | 50.0 | 66.7 | 42.9 | 28.6 | 66.7 | 78.6 | 66.7 | 76.9 | 50.0 | 25.0

7. Secondary Outcome: Crude Success Rate of Radiological Response to Treatment Evaluated by the Investigator at Day 42, Day 84 and EOT
Description: The Investigator evaluated radiological response to treatment at day 42, day 84 and EOT. Radiological response outcomes were described as Success [≥ 90% improvement,≥ 50% to < 90% improvement and ≥ 25% to < 50% improvement (for day 42 and EOT, if EOT occurs prior to day 42)]. End of treatment (EOT) is the last day of study drug administration, with an estimated duration up to 180 days.
Time Frame: Day 42, Day 84 and End of Treatment (EOT [Day 180])
Population: Modified Intent-To-Treat population (mITT)
Measure: Number; unit: percentage of participants
Arm/Group | mITT - Aspergillus [Renally Impaired] | mITT - Aspergillus [Not Renally Impaired] | mITT - Mucorales (Primary Therapy) | mITT - Mucorales (Refractory) | mITT - Mucorales (Intolerant) | mITT- Other Filamentous Fungi | mITT- Other Mould Species Only | mITT- Other Dimorphic Fungi | mITT- Other Non-Candida Yeast | mITT-Other Mixed Infection
Number analyzed (Participants) | 20 | 4 | 21 | 11 | 5 | 17 | 7 | 29 | 11 | 15
percentage of participants
  Day 42 | 35.0 | 75.0 | 40.0 | 0 | 40.0 | 46.7 | 20.0 | 32.1 | 9.1 | 28.6
  Day 84 | 40.0 | 50.0 | 25.0 | 11.1 | 40.0 | 40.0 | 20.0 | 37.0 | 0 | 7.1
  End of Treatment (EOT) | 35.0 | 50.0 | 30.0 | 22.2 | 20.0 | 33.3 | 40.0 | 55.6 | 10.0 | 14.3

8. Secondary Outcome: All-cause Mortality Through Day 42 and Day 84
Description: All-cause Mortality was assessed through Day 42 and Day 84 and summarized for ITT population End of treatment (EOT) is the last day of study drug administration, with an estimated duration up to 180 days.
Time Frame: Baseline to End of Treatment (EOT [Day 180])
Population: Intent-To-Treat population (ITT)
Measure: Number; unit: percentage of participants
Groups:
- Renally Impaired: Renally Impaired (RI) population consisted of participants who had proven or probable IFD as determined by the DRC. Classification by the DRC was based on the type of pathogen which was found to be the cause of participant's IFD. Renal impairment was defined as yes for participants who had a baseline eGFR-MDRD < 60 mL/min/1.73 m^2, no for patients who had a baseline eGFR-MDRD ≥ 60 mL/min/1.73 m^2. Overall there were 24 participants in the mITT-Aspergillus population out of which 20 participants were classified as Renally Impaired (RI).
- Not Renally Impaired: Not Renally Impaired (NRI) population consisted of participants who had proven or probable IFD as determined by the DRC. Classification by the DRC was based on the type of pathogen which was found to be the cause of participant's IFD. The Aspergillus-mITT population was presented by renal status (Renally Impaired and Not Renally Impaired). Overall there were 24 participants in the mITT- Aspergillus population out of which 4 participants were classified as Not Renally Impaired (NRI).
Arm/Group | Renally Impaired | Not Renally Impaired
Number analyzed (Participants) | 59 | 87
percentage of participants
  All-cause Mortality Through Day 42 | 22.0 | 16.1
  All-cause Mortality Through Day 84 | 30.5 | 20.7

9. Secondary Outcome: Safety - Overall Number of TEAEs
Description: A Treatment Emergent Adverse Events (TEAE) is any adverse event that starts after the first administration of study drug until 28 days after the last dose of study drug.
Time Frame: From the first study drug administration until 28 days after the last dose of study drug
Population: The safety analysis set (SAF) consists of all enrolled participants who received at least one dose of study drug as this was a non-comparative open-label study
Measure: Number; unit: participants
Groups:
- Isavuconazole: Participants received Isavuconazole intravenous (IV) or per oral (PO) over period of 2 days, on days 1 and 2 three doses of 200 mg were administered every 8 hours for a total of six doses. From Day 3 to End of Treatment (EOT) maintenance dose of 200 mg isavuconazole was administered once daily up to 180 days; with an option for extended treatment under specified criteria.
Arm/Group | Isavuconazole
Number analyzed (Participants) | 146
participants
  TEAEs | 139
  Study Drug-Related TEAEs | 60
  Serious TEAEs | 89
  Study Drug-Related Serious TEAEs | 13
  TEAEs Leading to Permanent Discontinuation of Stud | 19
  Study Drug TEAEs Leading to Perm Discontinuation | 7
  TEAEs Leading to Death | 44
  Study Drug-Related TEAEs Leading to Death | 1
  Deaths | 47
  Deaths Through 28 Days after Last Dose Study Drug | 42

ADVERSE EVENTS:
Time Frame: From the first administration of study drug until 28 days after the last dose of study drug. For the days when IV and oral doses were administered on the same day, the day was split into one-half day for each route's duration.
Description: The safety analysis set is identical to the intent -to-treat (ITT) population (i.e., all enrolled participants who received at least one dose of study drug) as this was a non-comparative open-label study.
Groups:
- Renally Impaired (RI): Renal impairment was defined as yes for participants who have a baseline as eGFR < 60 mL/min/1.73 m^2 by the Modification of Diet in Renal Disease (MDRD) formula.
- Not Renally Impaired (NRI): Not Renally impaired participants were defined as no if they have a baseline eGFR-MDRD ≥ 60 mL/min/1.73 m^2 by the Modification of Diet in Renal Disease (MDRD) formula.
Arm/Group | Renally Impaired (RI) | Not Renally Impaired (NRI)
Serious Adverse Events (participants affected / at risk) | 43/59 | 46/87
Other Adverse Events (participants affected / at risk) | 54/59 | 68/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Renally Impaired (RI) (N=59) | Not Renally Impaired (NRI) (N=87)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Electromechanical dissociation (Cardiac disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4
Death (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Cholangiolitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Acute graft versus host disease (Immune system disorders) | 2 | 0
Graft versus host disease (Immune system disorders) | 1 | 1
Lung transplant rejection (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Aspergillosis (Infections and infestations) | 1 | 2
BK virus infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 3 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 1 | 0
Bronchiectasis (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cytomegalovirus enteritis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 1
Empyema (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Fungal sepsis (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Mucormycosis (Infections and infestations) | 0 | 2
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 6
Pneumonia bacterial (Infections and infestations) | 1 | 2
Pneumonia blastomyces (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 2
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 2
Pseudomonas bronchitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 6 | 0
Sinusitis (Infections and infestations) | 1 | 0
Sinusitis fungal (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0
Zygomycosis (Infections and infestations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Aphasia (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 2
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 6 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arteritis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 0
Leukaemic infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Renally Impaired (RI) (N=59) | Not Renally Impaired (NRI) (N=87)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 6 | 2
Atrial fibrillation (Cardiac disorders) | 4 | 1
Sinus tachycardia (Cardiac disorders) | 3 | 2
Tachycardia (Cardiac disorders) | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 7 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 5 | 10
Diarrhoea (Gastrointestinal disorders) | 16 | 10
Haematochezia (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 19 | 14
Stomatitis (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 16 | 17
Asthenia (General disorders) | 1 | 7
Chills (General disorders) | 5 | 3
Fatigue (General disorders) | 4 | 2
Oedema peripheral (General disorders) | 8 | 8
Pain (General disorders) | 3 | 2
Pyrexia (General disorders) | 9 | 15
Clostridial infection (Infections and infestations) | 3 | 0
Clostridium difficile colitis (Infections and infestations) | 3 | 1
Herpes zoster (Infections and infestations) | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 5 | 6
Urinary tract infection (Infections and infestations) | 7 | 2
Blood alkaline phosphatase increased (Investigations) | 3 | 2
Gamma-glutamyltransferase increased (Investigations) | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 4 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 4
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3
Dizziness (Nervous system disorders) | 3 | 5
Headache (Nervous system disorders) | 11 | 14
Confusional state (Psychiatric disorders) | 7 | 2
Insomnia (Psychiatric disorders) | 5 | 8
Oliguria (Renal and urinary disorders) | 3 | 0
Renal impairment (Renal and urinary disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 7
Hypertension (Vascular disorders) | 3 | 5
Hypotension (Vascular disorders) | 5 | 5

LIMITATIONS AND CAVEATS:
Enrollment in the clinical study was suspended in January 2009 pending further characterization of newly identified impurities. After successful study completion resumption of enrollment started in April 2011 for the 9766-CL-0103/WSA-CS-003 study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication. At least sixty (60) days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy of all such manuscripts and materials , and allow Sponsor sixty (60) days to review and comment on them.